CLINICAL TRIAL: NCT02334046
Title: Effect-site Concentration of Remifentanil for Preventing Cough During Emergence in Elderly Patients
Brief Title: Remifentanil for Smooth Emergence in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AJIRB-MED-CT4-14-383
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Drug Usage
Keywords: tracheal extubation; remifentanil
MeSH Terms: interventions — Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elderly (Experimental): Remifentanil was maintained at predetermined effect-site concentration during the emergence period in elderly patients.
  Interventions: Drug: Remifentanil; Drug: Sevoflurane
- Adult (Active Comparator): Remifentanil was maintained at predetermined effect-site concentration during the emergence period in adult patients.
  Interventions: Drug: Remifentanil; Drug: Sevoflurane

INTERVENTIONS:
Drug: Remifentanil — Remifentanil was maintained at predetermined effect-site concentration during the periextubation period (initial concentration: 1.8 ng/ml) in elderly patients (65-80 years) .
  Other Names: Ultiva
  Arms: Adult
Drug: Remifentanil — Remifentanil was maintained at predetermined effect-site concentration during the periextubation period (initial concentration: 1.8 ng/ml) in adult patients (20-60 years) .
  Other Names: Ultiva
  Arms: Elderly
Drug: Sevoflurane — Anesthesia was maintained with sevoflurane with 1.5-2.0 vol% in air/50%oxygen mixture, and sevoflurane was adjusted to about 1.0 vol% 10 min before end of surgery.

SUMMARY:
Elderly patients show different pharmacokinetic and pharmacodynamic variables and usually need smaller doses of anaesthetic drugs than younger patients. The purpose of this study was to investigate the optimal effect-site concentration of remifentanil for preventing cough during emergence in elderly patients under sevoflurane and remifentanil anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II undergoing endoscopic sinus surgery or septoplasty under balanced anesthesia with sevoflurane and remifentanil

Exclusion Criteria:

* predicted difficult airway, body mass index > 30 kg/m2, history of obstructive sleep apnoea chronic respiratory disease or coughing, current smokers patients angiotensin converting enzyme-inhibitors

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of cough | from end of surgery to 5 min after tracheal extubation
  Number of cough or a strong and sudden contraction of the abdomen during periextubation periods

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeongki-do, South Korea